CLINICAL TRIAL: NCT06088277
Title: Texting in Community Health Center Dental Clinics to Reduce HIV Risk
Brief Title: Texting to Reduce Human Immunodeficiency Virus (HIV) Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-43228; UG3DE031249 (NIH)
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections
Keywords: Dental patients; Community Health Center Dental Clinics; Text messaging; HIV negative; HIV testing
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV text messages (TM HIV) (Experimental): Eligible participants randomized into this arm will receive text messages to reduce the risk for HIV and promote HIV testing.
  Interventions: Behavioral: TM HIV
- TM HL (Active Comparator): Eligible participants randomized into this arm will receive text messages to promote healthy living, but not specific to HIV risk or testing..
  Interventions: Behavioral: TM HL

INTERVENTIONS:
Behavioral: TM HIV — Participants will receive 5 intervention text messages (TM) about HIV risk and testing per week for the first 3 months and 3 messages per week for the last 3 months of the intervention.
  Arms: HIV text messages (TM HIV)
Behavioral: TM HL — Participants will receive 5 intervention text messages (TM) about promoting healthy living (HL) per week for the first 3 months and 3 messages per week for the last 3 months of the intervention.
  Arms: TM HL

SUMMARY:
This is a 3-year study to test the efficacy of a text message-based intervention program. Dental patients at 4 community health centers (n= 266) will be randomized to receive either text messages (TMs) regarding HIV prevention or TMs regarding overall wellness. Prior to enrolling the 266 participants, the investigators will conduct a feasibility pilot (n=20) to test the TM delivery as well as all study procedures. For both the pilot and the randomized clinical trial (RCT), recruitment will be conducted at 4 Community Health Center dental clinics (Codman Square, East Boston (both East Boston and South End locations), Geiger Gibson, and Upham's Community Health Centers). Recruitment materials (flyers and permission to contact forms) may also be made available at other clinics within the health centers.

The study will enroll English and Spanish-speaking patients who have at least one risk factor for HIV but are HIV-negative. Patients enrolled in the pilot will complete self-report surveys at baseline, 1 and 2 months. Participants enrolled in the RCT will complete self-report surveys baseline, 3, 6, and 12 months after baseline; receive and respond to TM assessments during the 6-month intervention.

ELIGIBILITY:
Inclusion Criteria:

* Give informed consent and document consent via a signed and dated informed consent form in REDCap
* Willing to comply with all study procedures and be available for the duration of the study
* Be able to read either in English or Spanish
* Be a dental clinic patient of record at one of our participating community health centers
* Has at least one risk factor for HIV defined as self-report of at least one of the following: Men who have sex with men; multiple sex partners, or intravenous drug use

Exclusion Criteria:

* Self-report of having HIV infection
* Participating in another HIV study or another text message study
* A woman who reports having sex exclusively with women
* Does not have a mobile phone or other device which can receive text messages from Agile Health
* Does not have unlimited texting on their mobile plan
* Has not used any type of text messaging at least once in the past month
* Single item literacy screening score of 2 or below.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2027-04-14 (Estimated); Study Completion 2027-04-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants that obtain HIV testing | 12 months
  The total number of participants that obtain HIV testing will be assessed from answers to a question in a study questionnaire.

SECONDARY OUTCOMES:
Adherence to pre-exposure prophylaxis (PrEP) | baseline, 3 months, 6 months, 12 months
  Participants will be asked to complete a study questionnaire where they will be asked if they adhered to PrEP.
PrEp Uptake | 3 months, 6 months, 12 months
  Percentage of participants who started PrEP since the last assessment
Condom use | 3 months, 6 months, 12 months
  Percentage of participants who used condoms consistently within the last month or at their last sexual encounter since the start of the intervention.
Intravenous Drug Use (IDU) | 3 months, 6 months, 12 months
  Among participants reporting IDU, percentage of participants who report using clean needles since the start of the intervention
Self-efficacy score | 6 months, 12 months
  This outcome will be assessed using a one-item measure with a 5-point Likert scale where: 1 = "Not at all", 2 = "Somewhat", 3 = "Undecided", 4 = "Not really", and 5 = "Very much". HIgher scores are more favorable.
Motivation to perform behaviours that reduce HIV risk | 3 months, 6 months, 12 months
  This outcome will be assessed using a one-item measure with a 5-point Likert scale where: 1 = "Not at all", 2 = "Somewhat", 3 = "Undecided", 4 = "Not really", and 5 = "Very much". HIgher scores are more favorable.
Outcome expectations regarding behaviors to reduce HIV risk. | 3 months, 6 months, 12 months
  This outcome will be assessed using a one-item measure with a 5-point Likert scale where: 1 = "Not at all", 2 = "Somewhat", 3 = "Undecided", 4 = "Not really", and 5 = "Very much". HIgher scores are more favorable.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Henshaw, DDS, MPH, Principal Investigator — Boston University Goldman School of Dental Medicine
Locations (2):
- United States (2):
  - South End Community Health Center, Boston, Massachusetts
  - East Boston Neighborhood Health Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT06088277/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT06088277/ICF_001.pdf